CLINICAL TRIAL: NCT06494891
Title: Translational Underpinnings of Motivation for Alcohol in Humans
Brief Title: Motivation for IV Alcohol Self-Administration in Humans
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Lara Ray, PhD, Professor, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: #23-000434; 1R01AA029701-01 (NIH)
Record Dates: First submitted 2024-07-02; First posted 2024-07-10 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism | interventions — Ethanol

STUDY DESIGN:
Intervention Model Description: All participants will receive intravenous alcohol.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Intravenous Alcohol (Experimental): Participants will receive 6% ethanol v/v in saline administered intravenously through the physiologically based pharmacokinetic model implemented in the Computerized Alcohol Infusion System.
  Interventions: Drug: Intravenous Alcohol

INTERVENTIONS:
Drug: Intravenous Alcohol — Participants will receive intravenous alcohol (6% ethanol v/v in saline; obtained from the Ronald Reagan UCLA Medical Center Investigational Drug Service) over the course of an alcohol challenge. During the challenge, participants will be administered alcohol designed to reach target BrACs of 20, 40, and 60 mg%, each over 15 min. After reaching the last target BrAC (0.06 g/dl) participants will complete a self-administration (SA) paradigm. Participants will be invited to work (button press) for alcohol according to a log-linear progressive ratio schedule.

SUMMARY:
The goal of this translational study is to understand different reasons why people between the ages of 21 and 65 with alcohol use disorder are motivated to self-administer alcohol. The main questions it aims to answer are:

* How does a person's desire for a reward affect their motivation to self-administer alcohol?
* How does a person's emotions affect their motivation to self-administer alcohol?
* How does a person's cognitive functioning affect their motivation to self-administer alcohol?

Participants will be asked to complete questionnaires about their mood, habits, and functioning and will complete an IV alcohol administration that will include pressing a button to receive additional doses of IV alcohol.

DETAILED DESCRIPTION:
This study combines alcohol challenge and progressive ratio self-administration methodologies to test the effects of each of the three dimensions of the Addictions Neuroclinical Assessment (ANA) on motivation for alcohol use. The experimental design consists of a translational study in which 210 individuals with current AUD (mild-to-severe) will complete an intravenous (IV) alcohol administration followed by a progressive ratio self-administration paradigm, where participants must press a button a number of times to receive an infusion of alcohol. All participants will be phenotyped for the three dimensions of the ANA, including incentive salience, negative emotionality, and executive dysfunction. For these models, the primary outcome in the progressive ratio self-administration paradigm will be: (a) breakpoint (i.e., the point in the progressive ratio model at which the participant stops button presses for alcohol) and (b) peak BrAC (i.e., the highest level of BrAC reached in the trial). At baseline and after the target BrAC of 0.06 g/dl in the alcohol challenge component of the paradigm, participants will report on (a) alcohol craving, (b) negative mood, and (c) loss of control over drinking. All participants will provide blood samples at baseline and at target BrAC =0.06 g/dl for analyses of the proposed exploratory biomarkers of HPA axis activation (ACTH, cortisol) and inflammation (IL-6, IL-10, TNF-α, CRP). The successful completion of this project will advance translational science of AUD by testing the ANA framework within a conceptually rich and valid translational task of motivation for alcohol in humans. Advanced data analytic methods (i.e., machine learning) and careful attention to AUD severity as a marker to AUD stage, will result in clinically useful findings that can inform AUD assessment, treatment, and biomarker development.

ELIGIBILITY:
Inclusion Criteria:

To be included in the study, participants must:

1. Be between the ages of 21 and 65
2. Have self-reported alcohol use in the past 30 days
3. Meet current (i.e., past 12 months) DSM-5 diagnostic criteria for alcohol use disorder mild-to-severe

Exclusion Criteria:

To be included in the study, participants must not:

1. Currently be treatment seeking, in treatment for alcohol use, or have a history of treatment in the 30 days prior to consent
2. Have current (last 12 months) DSM-5 diagnosis of substance use disorder for any psychoactive substances other than alcohol and nicotine
3. Have a lifetime DSM-5 diagnosis of schizophrenia, bipolar disorder, or any other psychotic disorder
4. Have current suicidal ideation or lifetime history of suicide attempt as reported on the Columbia-Suicide Severity Rating Scale (C-SSRS)
5. Have a positive urine screen for drugs other than cannabis
6. Be pregnant, nursing, or planning to become pregnant while taking part in the study; and must agree to one of the following methods of birth control (if female), unless she or partner are surgically sterile:

   * Oral contraceptives
   * Contraceptive sponge
   * Patch
   * Double barrier
   * Intrauterine contraceptive device
   * Etonogestrel implant
   * Medroxyprogesterone acetate contraceptive injection
   * Hormonal vaginal contraceptive ring
   * Complete abstinence from sexual intercourse
7. Have clinically significant abnormalities identified in the physical exam that may interfere with safe study participation (e.g. unstable cardiac, renal, or liver disease; diabetes; uncontrolled hypertension; or HIV)
8. Exceed Grade 2 laboratory abnormalities, based on FDA Guidance Document "Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials"
9. Currently use any medications known to interact with alcohol, including: antidepressants, anticonvulsants, opioids, benzodiazepines, medications for diabetes, and medications that affect alcohol metabolism
10. Have an intense fear of needles or have had adverse reactions to needle puncture
11. Have any other circumstances that, in the opinion of the investigators, would not be a good fit for study participation

Exclusion Criteria for Experimental Visit

To participate in the IV alcohol administration, participants must not:

1. Have a BrAC > 0.000 g/dl
2. Have clinically significant alcohol withdrawal symptoms as indicated by a score ≥ 10 on the Clinical Institute Withdrawal Assessment for Alcohol-Revised (CIWA-R)
3. Exceed Grade 2 clinical vital sign abnormalities, based on FDA Guidance Document "Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials"

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2024-01-16 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Incentive Salience, Craving, and Self-Administration | 10 hours
  Scores on the incentive salience factor of the ANA will correlate with craving during the challenge and self-administration during the progressive ratio.
Negative Emotionality, Negative Mood, and Self-Administration | 10 hours
  Scores on the negative emotionality factor of the ANA will correlate with relief from negative mood during the challenge and self-administration during the progressive ratio.
Executive Dysfunction, Loss of Control, and Self-Administration | 10 hours
  Scores on the executive dysfunction factor of the ANA will correlate with loss of control during the challenge and self-administration during the progressive ratio.

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No
Deidentified data will be uploaded to the National Institute on Alcohol Abuse and Alcoholism Data Archive.